CLINICAL TRIAL: NCT07249112
Title: DEFINIZIONE DEL PANORAMA GENOMICO DELLA MASLD (DEFINING THE GENOMIC LANDSCAPE OF METABOLIC STEATOTIC LIVER DISEASE)
Brief Title: DEFINITION OF THE GENOMIC LANDSCAPE OF MASLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Principal Investigation, Medical Doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DETECTIVE
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis; MASLD
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced MASLD Patients and Metabolic Controls (Experimental): This study aims to identify inherited genetic variants and somatic mutations associated with the progression of advanced Metabolic Dysfunction-Associated Steatotic Liver Disease MASLD.The research utilizes two distinct and extensively characterized cohorts for Whole-Genome Sequencing WGS analysis:
  * MASLD Cohort: Consists of 800 patients whose peripheral blood will undergo WGS at 20x coverage.
  * Metabolic Controls} Cohort: Comprises 2000 individuals matched for sex and metabolic risk factors who meet at least two criteria for metabolic syndrome but are free of MASLD. Their peripheral blood DNA will also be sequenced.
  Interventions: Other: genetic and somatic variants involved in its progression toward advanced fibrosis and hepatocellular carcinoma

INTERVENTIONS:
Other: genetic and somatic variants involved in its progression toward advanced fibrosis and hepatocellular carcinoma — The focusing is the attention on the genetic and somatic variants involved in its progression toward advanced fibrosis and hepatocellular carcinoma. Through Whole-Genome Sequencing WGS of 800 patients with advanced MASLD, 80 liver tissue samples, and 2000 controls, the study aims to:
  * Identify rare and structural genetic variants associated with the disease
  * Analyze the role of clonal hematopoiesis of indeterminate potential CHIP in MASLD progression.
  * Develop polygenic risk scores to improve risk stratification.

SUMMARY:
The Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is a leading cause of chronic liver disease globally, with a prevalence exceeding 30% in the population. MASLD is strictly associated with insulin resistance and cardiometabolic conditions, and in 20-30% of cases, it can progress to steatohepatitis (MASH), which is characterized by progressive liver damage and inflammation. In patients at higher risk, the disease can lead to the onset of advanced fibrosis, cirrhosis, and hepatocellular carcinoma (HCC). One of the main problems in the clinical management of MASLD is the absence of specific risk biomarkers and the lack of effective treatments, especially for patients with advanced-stage disease.

MASLD has a well-documented and enormous genetic component, with studies having identified several common variants associated with this pathology, such as those in the PNPLA3, TM6SF2, and MBOAT7 genes. However, these variants identified so far only explain a small part of MASLD's heritability, suggesting the contribution of rare loss-of-function (LoF) variants as well. Furthermore, scientific evidence indicates that the accumulation of somatic variants, both in hepatocytes and myeloid cells, could also play a key role in MASLD progression. In particular, clonal hematopoiesis of indeterminate potential (CHIP), which is a condition characterized by the presence of hematopoietic clones with somatic mutations often associated with leukemia and cardiovascular diseases, might favor the onset of hepatocellular carcinoma. However, the evidence available to date is still limited and requires further investigation and studies on larger cohorts.

The current study therefore aims to deepen this aspect through the analysis of the genetic profile using a Whole-Genome Sequencing (WGS) approach. DNA samples from peripheral blood from patients with advanced MASLD and peripheral blood DNA samples from controls presenting various associated metabolic risk factors will be sequenced.

In addition, 80 liver tissue samples from patients with advanced MASLD will also be sequenced to identify specific somatic mutations. The expected results from this study include the identification of new genetic variants associated with MASLD progression, the improvement of risk stratification through the development of polygenic risk scores, and the identification of potential therapeutic targets. This study represents a fundamental step for understanding the biology of MASLD and could have important clinical implications for disease management.

ELIGIBILITY:
Inclusion Criteria:

Specific Inclusion Criteria for Patients with Advanced MASLD:

* Patients with advanced MASLD defined as liver fibrosis ≥2 and/or the development of HCC (Hepatocellular Carcinoma);
* Patients enrolled in the context of the SERENA study and, where applicable, also in the context of the REASON study;
* Liver biopsy for suspected Non-Alcoholic Steatohepatitis (NASH) at the time of diagnosis;
* Cholecystectomies;
* Age [40-70 years];
* Patients who have signed the informed consent form.

Specific Inclusion Criteria for the Control Group:

Blood donors participating in the Liver Bible study aged between 40 and 70 years who are overweight or obese and have at least two of the following risk factors:

* Impaired fasting glucose or Diabetes Mellitus
* Dyslipidemia
* Arterial hypertension.

Exclusion Criteria:

Specific exclusion Criteria for Patients with Advanced MASLD:

* Positivity for chronic viral hepatitis (HCV-RNA and/or HBsAg);
* Positivity for other liver diseases such as autoimmune and viral hepatitis (Hepatitis B and C), hereditary hemochromatosis, alpha-1-antitrypsin deficiency, or Wilson's disease.

Specific Exclusion Criteria for the Control Group:

Subjects with chronic degenerative diseases will be excluded, with the exception of well-controlled hypertension and Type 2 Diabetes Mellitus that does not require pharmacological therapy (as is already standard practice for blood donation eligibility). Also excluded are donors aged > 65 and < 40 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2880 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Identifying Genetic Risk for Advanced MASLD | 11 months
  The study's outcome measures are defined by two distinct, primary endpoints. The first is the Number of Genetic Variants Associated with Advanced MASLD, reported as the total count of genetic variants (germline and/o somatic) exhibiting a statistically significant association with the risk of developing advanced Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD), defined as fibrosis ≥ 2 and/or hepatocellular carcinoma. The unit of measure for this outcome is Count (Number of variants). The second measure is the Odds Ratio (OR) for Association Between Germline Variants and Advanced MASLD, calculated by comparing the presence of specific germline variants in cases versus controls to determine the strength of their association with advanced MASLD.

SECONDARY OUTCOMES:
Mechanisms, Risk Stratification, and Therapy | 11 months
  This study aims to identify inherited genetic variants and somatic mutations associated with the progression of Advanced Metabolic Dysfunction-Associated Steatotic Liver Disease MASLD), utilizing two distinct and extensively characterized cohorts for Whole-Genome Sequencing (WGS) analysis:
  1. MASLD Cohort: Peripheral blood will undergo WGS text. A subset of 80 pathological liver tissue samples from 35 patients HCC/advanced fibrosis) will be sequenced at to identify somatic mutations.
  2. Metabolic Controls Cohort: Individuals with metabolic risk factors but lacking advanced MASLD; peripheral blood will be sequenced (WGS 20x). This cohort is deeply characterized, including OMICs data.
  The study's goals are to:
  * Identify genetic factors contributing to MASLD and HCC risk.
  * Develop polygenic risk scores (PRS) for better risk stratification.
  * Identify potential therapeutic targets for precision medicine in advanced MASLD.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT07249112/Prot_000.pdf